CLINICAL TRIAL: NCT04183049
Title: Improved Rehabilitation After Spinal Surgery in Adolescents: Prospective Observational Epidemiological Study of a Protocol Without Opioid
Brief Title: Improved Rehabilitation After Spinal Surgery in Adolescents
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC19_0255
Record Dates: First submitted 2019-11-14; First posted 2019-12-03 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative; Pain; Scoliosis; Spinal Fusion
Keywords: Dexmedetomidine; Analgesics; Opioid free anesthesia; Chronic postsurgical pain
MeSH Terms: conditions — Pain, Postoperative; Pain; Scoliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Impact of the OFA technique on postoperative recovery from adolescent spine surgery and the incidence of chronic postoperative pain.

DETAILED DESCRIPTION:
RACAROFA is an observational, prospective study based on the hypothesis that the OFA technique effectively improves the long-term postoperative rehabilitation of adolescents and reduces the incidence of CPSP. A prospective French multicentre study on this topic is currently not feasible, as other multicentre studies (pain monitoring by the ANI, blood saving strategy) would interfere with potential recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patent with idiopathic or secondary surgical scoliosis
* Management by the paediatric anaesthesia team at the Mother and Child - Hospital of the University Hospital of Nantes
* Non-opposition to inclusion in the study collected orally from the patient and parents
* Satisfying oral and written comprehension of the French language, without interpreter
* Ability to participate in a telephone interview

Exclusion Criteria:

* Patient that does not understand French correctly
* Patient unable to express himself/herself correctly in French
* Patient with a non-scoliotic surgical spinal pathology
* Refusal to participate in the study
* Absence of a record of non-opposition to participation in the study from the patient and his or her parents
* Cerebral palsy or any other condition that does not allow participation in a telephone interview without particular difficulty.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - As the study concerns a specifically paediatric pathology, minors will not be excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic postsurgical pain after surgery in the adolescent cohort included in the study RACAROFA | Three months after surgery
  Pain at the surgical site, rated at more than 3 on a numerical scale graduated from 0 (no pain) to 10 (maximum pain) during a telephone interview.
Incidence of chronic postsurgical pain after surgery in the adolescent cohort included in the study RACAROFA | Sixth months after surgery
  Pain at the surgical site, rated at more than 3 on a numerical scale graduated from 0 (no pain) to 10 (maximum pain) during a telephone interview.

SECONDARY OUTCOMES:
Occurence of a postoperative opioid-related adverse event | Within the first 48 hours after extubation
  postoperative hypoxemia or PONV (postoperative nausea and vomiting) or excessive sedation. Postoperative hypoxemia is defined as an oxygen saturation (SpO2) < 95% with a need for oxygen supplementation within the first 48h after extubation.
  PONV is defined by use of antiemetics of PONV within the first 48h after extubation.
  Excessive sedation is defined by a score of 3 in a scale of sedation wich is S1 awake, S2 mild drowsiness, S3 non awakenable.
Level of preoperative quality of life | Three month after surgery
  SRS-30 score (Scoliosis Research Society Health-Related Quality of Life Questionnaire), during a telephone interview. Score between 1 and 5 where 5 is the higher level of quality of live.
Postoperative opioid consumption | Within the 2 first weeks postsurgery
  Cumulative consumption of opioid in mg/kg.
Level of preoperative quality of life: SRS-30 score | Sixth month after surgery
  SRS-30 score (Scoliosis Research Society Health-Related Quality of Life Questionnaire), during a telephone interview. Score between 1 and 5 where 5 is the higher level of quality of live.
Postoperative rehabilitation | Within the first 2 weeks postsurgery
  Number of days between surgery and first deambulation
Length of stay in the hospital | Within the first 2 weeks postsurgery
  Number of days in the hospital.
Level of preoperative and postoperative anxiety in the adolescent cohort included in the study RACAROFA | Two weeks before surgery
  State trait anxiety Inventory for Children (STAIC) score evaluated during a telephone interview. Score between 20 and 60, where 60 is the higher level of anxiety
Level of preoperative and postoperative anxiety in the adolescent cohort included in the study RACAROFA | three months after surgery
  State trait anxiety Inventory for Children (STAIC) score evaluated during a telephone interview. Score between 20 and 60, where 60 is the higher level of anxiety
Level of preoperative and postoperative anxiety in the adolescent cohort included in the study RACAROFA | sixth months after surgery
  State trait anxiety Inventory for Children (STAIC) score evaluated during a telephone interview. Score between 20 and 60, where 60 is the higher level of anxiety
Incidence of postoperative neuropathic pain in the adolescent cohort included in the study RACAROFA. | Three months after surgery
  Modified DN4 score superior at 4.
Incidence of postoperative neuropathic pain in the adolescent cohort included in the study RACAROFA. | Six months after surgery
  Modified DN4 score superior at 4.
Postoperative antalgics consumption other than opioid | Within the first 2 weeks postsurgery
  Cumulative antalgics consumption other than opioid.
Incidence of preoperative pain in the adolescent cohort included in the study RACAROFA. | Two weeks before surgery
  Back pain, rated at more than 3 on a numerical scale graduated from 0 (no pain) to 10 (maximum pain) during a telephone interview.
Level of preoperative and postoperative catastrophism in the adolescent cohort included in the study RACAROFA. | Two weeks before surgery, three and sixth months after surgery
  Pain castrophizing scale for adolescent, score evaluated during a telephone interview. Score between 0 and 52, where 52 is the higher level of catastrophism.
Level of preoperative and postoperative catastrophism in the adolescent cohort included in the study RACAROFA. | three months after surgery
  Pain castrophizing scale for adolescent, score evaluated during a telephone interview. Score between 0 and 52, where 52 is the higher level of catastrophism.
Level of preoperative and postoperative catastrophism in the adolescent cohort included in the study RACAROFA. | sixth months after surgery
  Pain castrophizing scale for adolescent, score evaluated during a telephone interview. Score between 0 and 52, where 52 is the higher level of catastrophism.
Level of preoperative and postoperative catastrophism in one of the parents of each adolescent included in the study RACAROFA. | Two weeks before surgery, three and sixth months after surgery
  Pain castrophizing scale for adult, score evaluated during a telephone interview. Score between 0 and 52, where 52 is the higher level of catastrophism.
Level of preoperative and postoperative catastrophism in one of the parents of each adolescent included in the study RACAROFA. | three months after surgery
  Pain castrophizing scale for adult, score evaluated during a telephone interview. Score between 0 and 52, where 52 is the higher level of catastrophism.
Level of preoperative and postoperative catastrophism in one of the parents of each adolescent included in the study RACAROFA. | sixth months after surgery
  Pain castrophizing scale for adult, score evaluated during a telephone interview. Score between 0 and 52, where 52 is the higher level of catastrophism.
Level of preoperative quality of life. | Two weeks before surgery
  SRS-22 score (Scoliosis Research Society Health-Related Quality of Life Questionnaire), during a telephone interview. Score between 1 and 5 where 5 is the higher level of quality of live

CONTACTS AND LOCATIONS:
Overall Officials: Corine LEJUS, PUPH, Principal Investigator — Nantes University Hospital; Guy LETELLIER, PH, Principal Investigator — Establishment for Children and Adolescents in the Nantes Region
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France